CLINICAL TRIAL: NCT05433805
Title: Prospective Evaluation of Lifestyle-modifying Interventions on Disease Parameters, Inflammatory and Metabolic Processes in Low-risk MDS Patients
Brief Title: Lifestyle-modifying Interventions in Low-risk MDS Patients
Acronym: MDS-LIME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020
Record Dates: First submitted 2022-05-23; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndrome; fasting-mimicking diet; physiotherapy; lifestyle modification; inflammation; metabolism
MeSH Terms: conditions — Myelodysplastic Syndromes; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMD first (Experimental): Patients receive nutritional counselling on the principles of the FMD diet and individual recommendations for optimising the micronutrient balance (vitamins, trace elements) based on their corresponding baseline values. A food diary is given to the patients to assess treatment adherence on FMD days.
  This is followed by a combined nutritive and physiotherapeutic interventions from week 13 for a further 3 months. Patients will be instructed about ambulatory exercises during a physiotherapeutic counselling, scheduled in week 13. Physiotherapy exercises should only be carried out on FMD-free days. Patients also receive a diary in which they document daily physical activity.
  Interventions: Other: Fasting-mimicking diet (FMD) and physiotherapy
- Physiotherapy first (Experimental): Patients receive physiotherapy counselling, with structured ambulatory exercises shown and explained. The patients receive a diary where they have to document their physical activity every day.
  This is followed by a combined nutritive and physiotherapeutic interventions from week 13 for a further 3 months. For this purposphe, nutritional counselling on the principles of the FMD diet is planned for week 13. In addition, individual recommendations for optimising the micronutrient balance (vitamins, trace elements) are given based on the respective baseline values. The physiotherapeutic exercises are to be carried out only on FMD-free days. Patients will also be given a food diary to assess treatment adherence on FMD days.
  Interventions: Other: Fasting-mimicking diet (FMD) and physiotherapy

INTERVENTIONS:
Other: Fasting-mimicking diet (FMD) and physiotherapy — FMD is a diet held monthly during five days with the restriction of calories to less than 1000 kcal, glucose and proteins.
  Physiotherapy will be organized as home-based exercises explained by the physiotherapeutist at the beginning of the study.

SUMMARY:
Myelodysplastic syndromes (MDS) are acquired clonal stem cell diseases characterized by hematopoietic cell dysplasia, cytopenia, and the risk of progression to acute myeloid leukemia. In addition to clonal changes in the hematopoietic stem and progenitor cells itself, growing evidence suggests that inflammatory and metabolic changes in the bone marrow microenvironment play an important role in disease development and maintenance of the malignant clone. The positive impact of dietary interventions (e.g. fasting) and physical activity on inflammation and metabolic parameters could be shown in various benign inflammatory disease entities (e.g. atherosclerosis, chronic renal insufficiency, cystic fibrosis etc.).

The aim of this study is to describe the hematological, metabolic, inflammatory, and microbiological changes after combined lifestyle-modifying interventions (outpatient physiotherapy and fasting mimicking diet (FMD) in patients with low-risk MDS.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age
2. Cytomorphologically confirmed MDS or MDS/MPN according to WHO criteria (incl. MDS-RARS-T, CMML)
3. IPSS-R very low, low, or intermediate
4. Hemoglobin <11 g/dL (6.8 mmol/l)
5. Non-transfusion dependent (NTD) per IWG 2018 criteria (≤2 blood transfusions within 16 weeks prior to inclusion in the study)
6. ECOG≤2
7. Body mass index (BMI) ≥ 20 kg/m2
8. Written informed consent of the subject after clarification

Exclusion Criteria:

1. AML
2. MDS IPSS-R high or very high
3. History of HSCT
4. MDS-specific drug therapy (including erythropoietin, erythropoiesis-modulating agents, lenalidomide, iron chelation, hypomethylating agents) ongoing or planned in the next 6 months
5. Diabetes mellitus requiring therapy or any other known metabolic disease
6. Application of systemic cortisone-containing drugs
7. Known psychiatric eating disorder (e.g. anorexia nervosa, bulimia)
8. Physical inability to follow the physical and/or nutritive interventions
9. simultaneous participation in another interventional clinical trial (including within the last 4 weeks before inclusion)
10. addictions or other illnesses that do not allow the person concerned to assess the nature and extent of the clinical trial and its possible consequences
11. pregnant or breastfeeding women
12. indications that the subject is unlikely to adhere to the protocol (e.g., lack of compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Hematological improvement | 24 weeks
  Hemoglobin level at the EOT visit, g/dL

SECONDARY OUTCOMES:
Evaluation of a priori metabolic parameters of MDS patients after combined physiotherapeutic and nutritive interventions | 6 months
  Panel measurement, mg/dL
Evaluation of a priori inflammatory parameters of MDS patients after combined physiotherapeutic and nutritive interventions | 6 months
  Panel measurement, ng/mL
Patients' adherence to therapy as an expression of the relevance of the lifestyle-modifying interventions in everyday life | 6 months
  Diary analysis
Impact on quality of life | 6 months
  QUALMS questionnaire
Impact on fatigue | 6 months
  Mean Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue score

IPD SHARING:
Plan to Share IPD: Undecided